CLINICAL TRIAL: NCT05460182
Title: Coronally Advanced Flap With and Without Connective Tissue Graft for the Treatment of Single Maxillary Gingival Recession With Loss of Inter-dental Attachment. A Randomized Controlled Clinical Trial - 10 Years Results
Brief Title: Treatment of Single Maxillary Gingival Recession With Loss of Inter-dental Attachment. A Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Dr. Francesco Cairo, Prof., University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RT2-10
Record Dates: First submitted 2022-07-06; First posted 2022-07-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two examiners, blinded with respect to the surgical procedures, assessed all the clinical and aesthetic outcomes of treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF+CTG (Experimental): After local anaesthesia, a split-full-split thickness flap was elevated. The papillae adjacent to the involved tooth were then de-epithelialized. A gentle root debridement was performed.
  A 1-2-mm-thick CTG was harvested using a single incision approach from the palate in the area between the second pre-molar and the second molar. The wound on the donor site of the palate was then sutured. The graft was positioned on the instrumented root surface immediately apical or at the level of the CEJ and then stabilized using a compressive crossing suture, anchored to the periosteum apical to the graft and closed with a palatal knot. The flap was coronally displaced 1-2 mm above the CEJ and sutured
  Interventions: Other: CAF+CTG
- CAF (Active Comparator): After local anaesthesia, a split-full-split thickness flap was elevated. The papillae adjacent to the involved tooth were then de-epithelialized. A gentle root debridement was performed. The flap was coronally displaced 1-2 mm above the CEJ and sutured
  Interventions: Other: CAF

INTERVENTIONS:
Other: CAF+CTG — Coronally Advanced Flap + Connective Tissue Graft
  Arms: CAF+CTG
Other: CAF — Coronally Advanced Flap
  Arms: CAF

SUMMARY:
Background: The aim of this randomized clinical trial (RCT) was to evaluate the adjunctive benefit of Connective Tissue Graft (CTG) to Coronally Advanced Flap (CAF) for the treatment of gingival recession associated with inter-dental clinical attachment loss equal or smaller to the buccal attachment loss (RT2). Material and Methods:The patients were randomly assigned to CAF+CTG (test group) or to CAF alone (Control group). Measurements were performed by a blind and calibrated examiner. Outcome measures included complete root coverage (CRC), recession reduction (RecRed), Root coverage Esthetic Score (RES), intra-operative and post-operative morbidity, and root sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Smoking < 20 cigarettes/day.
* Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) < 15% (measured at four sites per tooth).
* Presence of at least one RT2 (Cairo et al. 2011) buccal gingival recession > 2 mm of depth
* Only gingival recessions localized at upper central and lateral incisors, canine, and first and second pre-molars associated with aesthetic problems and/ordental hypersensitivity were considered.
* Presence of an identifiable CEJ

Exclusion Criteria:

* Systemic diseases or pregnancy.
* Systemic antibiotic therapy in the last 6 months.
* Active periodontal disease with sites showing probing depth >4 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Complete Root Coverage (CRC) | After the intervention (10 years)
  Complete Root Coverage: absence of gingival recession (Yes/No)

SECONDARY OUTCOMES:
Recession Reduction (RecRed) | After the intervention (10 years)
  Change of the gingival recession, in mm
Root Coverage Aesthetic Score (RES) | After the intervention (10 years)
  A scoring system ranging from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florence, Florence, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cairo F, Cortellini P, Barbato L, Masseti L, Mervelt J, Nieri M, Pini Prato GP, Tonetti MS. Long-term comparison of root coverage procedures at single RT2 maxillary gingival recessions: Ten-year extension results from a randomized, controlled clinical trial. J Clin Periodontol. 2023 Apr;50(4):511-519. doi: 10.1111/jcpe.13778. Epub 2023 Jan 24. PMID 36644804